CLINICAL TRIAL: NCT00145002
Title: Phase III Study of VCAP-AMP-VECP vs. Biweekly CHOP in Aggressive Adult T-cell Leukemia-lymphoma (ATLL): Japan Clinical Oncology Group Study, JCOG9801.
Brief Title: A Study for Aggressive Adult T-cell Leukemia-lymphoma (ATLL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Clinical Oncology Group (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG9801; C000000066
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Adult T-cell Leukemia; Lymphoma
Keywords: ATLL; chemotherapy; phase III study; VCAP-AMP-VECP; biweekly-CHOP
MeSH Terms: conditions — Leukemia-Lymphoma, Adult T-Cell; Lymphoma | interventions — Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: VCAP-AMP-VECP with G-CSF and intrathecal prophylaxis
Drug: biweekly-CHOP with G-CSF and intrathecal prophylaxis

SUMMARY:
To test the superiority of VCAP-AMP-VECP regimen over biweekly-CHOP in aggressive ATLL in terms of survival benefit.

DETAILED DESCRIPTION:
Nothing to describe.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ATL was made based on seropositivity for HTLV-I by either enzyme-linked immunosorbent assay or particle agglutination assay, and histologically- and/or cytologically-proven peripheral T-cell malignancy
2. Aggressive ATL, i.e., acute-, lymphoma- or unfavorable chronic-type ATL
3. Aged 15-69 years
4. No prior chemotherapy or radiotherapy
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-3 or 4 as a result of hypercalcemia
6. Preserved organ (bone marrow, liver, kidney, heart and lung) functions
7. All patients were required to provide written informed consent

Exclusion Criteria:

1. Diabetes mellitus necessitating treatment with insulin
2. Active systemic infection
3. Cardiac disorders expected to become worse as a result of the DOX-containing regimen
4. Acute hepatitis, chronic hepatitis or liver cirrhosis
5. Positive for HBs Ag or anti-HCV Ab
6. Active concurrent malignancy
7. Other serious medical or psychiatric conditions
8. Pregnancy or breast feeding
9. Central nervous system involvement by ATL cells

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130
Dates: Start 1998-08; Study Completion 2004-12

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Toxicity
CR rate
Progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Masao Tomonaga, MD, PhD, Study Chair — Nagasaki University Graduate School of Biomedical Science
Locations (1):
- Nagasaki University Graduate School of Biomedical Science, Nagasaki, Nagasaki, Japan

REFERENCES:
- See also: Related Info — http://www.jcog.jp/